CLINICAL TRIAL: NCT03160755
Title: Developing a Group-based Positive Psychology and Physical Activity Intervention in Patients With Metabolic Syndrome: Qualitative Research Phase
Brief Title: Motivation-Audit-Positive Psychology Intervention Study
Acronym: MAPP-I
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rachel Millstein, Assistant in Psychology, Massachusetts General Hospital
Other Study IDs: 2016P002824
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Qualitative Interviews: Adult outpatients with metabolic syndrome.

SUMMARY:
Specific Aim #1: To identify, through qualitative research, deficits in positive emotional states (e.g., positive affect, optimism) and associated barriers to completing health behaviors, like physical activity and healthy eating, in patients with metabolic syndrome (MetS).

Hypothesis: Participants will be able to complete semi-structured interviews, providing information about their positive emotional states, linking the presence of positive emotions to better adherence to health-related behaviors, and identifying additional barriers (e.g., logistic, motivational) to completing such behaviors.

DETAILED DESCRIPTION:
This qualitative interview study will focus on the development of a novel positive psychology (PP) and motivational interviewing (MI) intervention that is adapted for patients with MetS. For this phase, participants will be primary care patients recruited through Massachusetts General Hospital's research opt-in program (Research Options Direct to You [RODY]). We will complete phone interviews with patients (n=20) with MetS within two weeks of enrollment in the study.

In this project, we hope to do the following:

1. Identify, through qualitative research, deficits in positive emotional states in primary care patients with MetS.
2. Examine potential links between positive emotional deficits and impaired health behaviors (low physical activity, unhealthy dietary patterns), as well as links between positive emotional states and successful health behaviors.
3. Identify other barriers to health behavior completion, such as social support and neighborhood resources.
4. Explore strategies to enhance positive emotional states in MetS patients and inquire about the utility of potential PP exercises in these patients.
5. Ask participants for feedback about intervention delivery preferences (e.g., session length, time of day, duration of intervention).
6. Develop a preliminary PP-MI based group intervention using the above information.

ELIGIBILITY:
Inclusion Criteria:

* Both of the two MetS components most strongly related to MetS outcomes and most sensitive to lifestyle change:
* elevated abdominal obesity (waist circumference >102 cm in men or >88 cm in women)
* If waist circumference is not available, body mass index (BMI) will be used as a surrogate measure based on prior research (BMI ≥29.1 kg/m2 for men and 27.2 kg/m2 for women).

AND

* elevated blood pressure (systolic ≥130 and/or diastolic ≥85 mm Hg or be on blood pressure medication).
* Plus ≥1 additional MetS component:
* Serum triglycerides ≥150 mg/dL
* High-density lipoprotein (HDL) cholesterol <40 mg/dL in men or <50 mg/dL in women
* Fasting plasma glucose >100mg/dL.
* Suboptimal physical activity defined as <150 minutes/week moderate intensity activity, which represents less than national-level recommendations.

Exclusion Criteria:

* Inability to speak/read English
* Cognitive deficits impeding ability to participate or provide informed consent (measured by a 6-item screen)
* Illness likely to lead to death in the next 6 months per PCP
* Current treatment for cancer, liver, or renal disease
* Pregnancy
* Documented severe mental illness (e.g., psychosis, suicidality)
* No telephone access
* Inability to be physically active
* Diabetes or known or suggested cardiac disease, given that this is a primary prevention study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metabolic syndrome patients with a Partners Healthcare provider
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Qualitative Data | Baseline
  Themes related to: health behaviors, barriers to completing health behaviors, positive emotional/cognitive experiences and how these may impact adherence to the MetS health behaviors of interest (primarily physical activity).

SECONDARY OUTCOMES:
Dispositional Optimism | Baseline
  Measured by the Life Orientation Test-Revised (LOT-R)
Positive Affect | Baseline
  Measured using the 10 positive affect items on the Positive and Negative Affect Schedule (PANAS)
Anxiety | Baseline
  Measured by the anxiety subscale of the Hospital Anxiety and Depression Scale (HADS)
Depression | Baseline
  Measured by the depression subscale of the Hospital Anxiety and Depression Scale (HADS)
Environmental Barriers and Resources | Baseline
  Measured using the Neighborhood Environment Walkability Scale - Abbreviated (NEWS-A)
Barriers to Physical Activity | Baseline
  Measured using the Barriers to Being Active Quiz
Health Related Quality of Life | Baseline
  Assessed via the Medical Outcomes Study Short Form-12 (SF-12)
Physical Activity | Baseline
  Assessed using the well-validated International Physical Activity Questionnaire-Short Form (IPAQ-SF)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Millstein, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No